CLINICAL TRIAL: NCT06785545
Title: The Value of Urinary CA19-9 Level in the Differential Diagnosis of Neurogenic and Non-Neurogenic Lower Urinary Tract Dysfunction in Children
Brief Title: Urinary CA19-9 Level in the Differential Diagnosis of Neurogenic and Non-Neurogenic Lower Urinary Tract Dysfunction in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MAR.UAD.0014
Record Dates: First submitted 2024-12-23; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-01

CONDITIONS: Lower Urinary Track Symptoms
Keywords: ca19-9

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Control Group (Active Comparator): child with haven't lower urinary tract symptoms
  Interventions: Diagnostic Test: CA19-9
- Norogenic Lower Urinary Tract Symptoms Group (Active Comparator): child have lower urinary tract symptoms with neuroulogical etiology
  Interventions: Diagnostic Test: CA19-9
- Lower Urinary Tract Symptoms Group (Active Comparator): They haven't norogenic etiyology
  Interventions: Diagnostic Test: CA19-9

INTERVENTIONS:
Diagnostic Test: CA19-9 — All patients Ca19-9 levels calculated from their urinary samples

SUMMARY:
It has been shown in the literature that urinary CA19-9 levels are associated with the degree of hydronephrosis and the anteroposterior diameter of the renal pelvis. Additionally, this marker has been reported as a potential indicator of kidney damage related to obstructive uropathies. A study conducted in our clinic, which has yet to be published, investigated CA19-9 levels in children with hydronephrosis of different etiologies. It found a statistically significant difference in CA19-9 levels between children with neurogenic and non-neurogenic lower urinary tract (LUT) dysfunction (Evaluation of Spot Urine Carbohydrate Antigen 19-9, Sodium, Potassium, and Creatinine Levels as Biomarkers for Differential Diagnosis of Hydronephrosis and Detection of Kidney Damage in Children Aged 0-16: A Prospective Study, Kütükoğlu et al.). Based on this, the hypothesis was formulated that urinary CA19-9 might be a potential biomarker for indicating neurological deficits in children presenting with LUT symptoms. Therefore, this study aimed to compare CA19-9 levels in a larger group of children with neurogenic and non-neurogenic LUT dysfunction.

DETAILED DESCRIPTION:
A total of 25 children with non-neurogenic etiologies and 25 children with neurogenic etiologies who presented to our clinic with LUT dysfunction were prospectively included in the study. A control group of 15 healthy children was also included. Urine samples were collected from the children, centrifuged at 3000 rpm for 4 minutes, and stored at -25°C. Urinary CA19-9 was analyzed using ELISA, and creatinine levels were measured for configuration in the spot urine samples. Additionally, for the neurogenic group, scintigraphy, urinary ultrasonography, voiding cystourethrography, and urodynamic (UD) parameters were recorded. Children with active urinary tract infections, malignancy, or congenital urinary anomalies were excluded from the study. Urinary CA19-9 levels were compared between the groups, and subgroup analysis was performed within the neurogenic group based on urodynamic parameters and the presence of upper urinary tract (UUT) damage. The presence of vesicoureteral reflux, hydronephrosis, or renal scarring was considered as UUT damage.

ELIGIBILITY:
Inclusion Criteria:

* lower urinary tract symptoms
* <18 years old

Exclusion Criteria:

* active urinary tract infections
* malignancy
* congenital urinary anomalies

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Ca19-9 levels | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: CAGRI A. SEKERCİ, Study Director — MARMARA UNİVERSİTY SCHOOL OF MEDİCİNE DEPARTMENT OF UROLOGY
Locations (1):
- Marmara University School of Medicine Urology Department, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No